CLINICAL TRIAL: NCT05726253
Title: Supportive Treatment and Antibiotics for Mild Pediatric Pneumonia
Acronym: STAMPP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023-5696
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia; Pediatric Respiratory Diseases; Antibiotic Use; Community-acquired Pneumonia
Keywords: Pediatrics; Pediatric CAP; Pediatric Pneumonia; Antibiotic Use
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Palliative Care; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Pilot Feasibility Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Randomization to receive either oral placebo or amoxicillin for a standard course (7 days)
  Interventions: Drug: Supportive Care + Placebo (no antibiotics)
- Amoxicillin (Active Comparator): Randomization to receive either oral amoxicillin or placebo for a standard course (7 days)
  Interventions: Drug: Supportive Care + Amoxicillin

INTERVENTIONS:
Drug: Supportive Care + Amoxicillin — Participants will be randomized to receive oral amoxicillin for a standard course (7 days)
  Arms: Amoxicillin
Drug: Supportive Care + Placebo (no antibiotics) — Participants will be randomized to receive oral placebo for a standard course (7 days)
  Arms: Placebo

SUMMARY:
National guidelines make two recommendations for treatment of young children with mild pneumonia - one to avoid routine antibiotics and another to use narrow-spectrum antibiotics. No studies have compared the effectiveness of these two approaches. This pilot study will evaluate study processes and feasibility of a future clinical trial that proposes to test whether low-risk children managed as outpatients with mild community-acquired pneumonia (CAP) treated with supportive treatment without antibiotics will have a similar clinical response, with fewer adverse effects, compared with those treated with a supportive treatment plan that includes antibiotics.

DETAILED DESCRIPTION:
This pilot clinical trial is a randomized, placebo-controlled, double-blinded trial assessing the feasibility of comparing supportive care+amoxicillin to supportive care without antibiotics (i.e., placebo) in children 12 months to <6 years of age who present to the ED with community-acquired pneumonia (CAP) and who will be treated as outpatients.

This trial will enroll over a 6-month period and take place at Ann and Robert H. Lurie Children's Hospital of Chicago. Clinical research coordinators (CRCs) will screen for and enroll eligible children.

Through an online system, participants will be randomized to a 7-day course of either amoxicillin (80-100 mg/kg divided BID up to 4,000 mg/day) or matching placebo. All patients will receive a supportive care treatment bundle that includes antipyretics, honey, and saline spray, in addition to instructions on how to manage lower respiratory infections.

The guardians of participants will be asked to complete an online daily symptom diary during the first 6 days after the initial study visit. Participants will have daily telehealth evaluations by clinicians for the first three days after the index study visit. The primary outcome will be assessed at day 7, using telehealth technology. A final follow-up, performed by site research staff, by telephone call, will occur at Day 21 to assess overall disease course and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-71 months; and
2. Diagnosis of CAP, defined using established criteria:

   1. Signs and symptoms of lower respiratory tract infection (LRTI), defined as any of the following:

      * new or different cough; or
      * new or different sputum production; or
      * chest pain; or
      * dyspnea/shortness of breath; or
      * documented tachypnea; or
      * abnormal findings consistent with LRTI on physical examination (e.g., crackles/rales, rhonchi, wheezing) and
   2. Fever, defined as tactile temperature at home or measured temperature ≥38ºC rectal, ≥37.7ºC oral, or ≥37.5ºC axillary, and
   3. Clinician diagnosis of CAP,
3. Intention to treat as an outpatient after ED/primary care visit, and
4. Mild disease, defined as lack of respiratory distress per adapted Pediatric Infectious Diseases Society/Infectious Diseases Society of America criteria: none of the following: dyspnea, concerning retractions per treating clinician, grunting, nasal flaring, apnea, altered mental status, SpO2<93% in room air, or respiratory rate >50 breaths per minute for ages 12-24 months or respiratory rate > 40 breaths per minute if age>24 months.

Exclusion Criteria:

1. Hospitalization within one-month preceding study visit; or
2. Incomplete immunization status (<2 doses of Hib and pneumococcal vaccines); or
3. Chronic complex medical conditions (chronic heart disease followed by cardiology, chronic lung disease (not including asthma), congenital airway or lung malformations, cystic fibrosis, tracheostomy tube, requiring positive-pressure ventilation, neuromuscular disorders affecting the lungs or chest wall); or
4. Conditions that compromise the immune system (HIV with CD4 count less than 400, primary immunodeficiency, asplenia, sickle cell disease, receipt of hematopoietic stem cell or solid organ transplant, cancer on active chemotherapy, immunosuppressive agents, daily corticosteroids for more than 7 consecutive days in past 14 days); or
5. Systemic antibiotic receipt (more than 1 dose) within the previous two weeks of CAP diagnosis; or
6. Radiographic findings of a consolidation of a concerning size or complexity in the view of the treating clinician; or
7. Radiographic findings of complicated pneumonia (pleural effusion larger than trace in size, empyema, [complex/septated collection] abscess, necrotic lung disease); or
8. Pneumonia known to be due to bacterial source at the time of enrollment, as documented by blood culture or PCR if available, or another clear source of bacterial infection requiring immediate antibiotics; or
9. Diagnosed with pneumonia in the previous month; or
10. Provider diagnosis of aspiration pneumonia; or
11. Severe (type 1) drug allergy to amoxicillin; or
12. Any other condition that in the judgement of investigators or the clinical team could affect safety of the subject; or
13. No access to a telephone or video technology for follow-up; or
14. Current enrollment in another clinical trial of an investigational agent; or
15. Previous enrollment in this trial; or
16. Parent/guardian non-English or non-Spanish speaking; or
17. Known allergy to milk and/or red dye.

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate Per Month | Measured at completion of pilot trial (6 months)
  Total number of participants enrolled divided by the total number of active enrollment months

SECONDARY OUTCOMES:
Consent Rate | Measured at completion of pilot trial (6 months)
  Number of eligible participants approached regarding trial participation who provided informed consent to participate in the trial compared with number of participants approached for participation
Lost to Follow-Up at Day 7 | Measured at completion of pilot trial (6 months)
  Number of enrolled participants who did not complete the Day 7 follow-up visit
Lost to Follow-Up at Day 21 | Measured at completion of pilot trial (6 months)
  Number of enrolled participants who did not complete the Day 21 follow-up visit

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, a public use dataset will not be developed.